CLINICAL TRIAL: NCT04779008
Title: Long-term Remote Ischemic Preconditioning Improves Myocardial Perfusion and Prognosis of Patients After Coronary Artery Bypass Grafting
Brief Title: Long-term Remote Ischemic Preconditioning Improves Myocardial Perfusion and Prognosis of Patients After CABG
Acronym: L-RIPC-CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE202101
Record Dates: First submitted 2021-02-04; First posted 2021-03-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: Experimental Group 1:The patient underwent one RIPC (Four five-minute cycles of upper limb ischaemia and Four five-minute pauses using a blood pressure cuff air vehicle to 200 mmHg) 4 hours before surgery, then normal surgery, and RIPC was performed on the second day after surgery and every day after surgery, which lasted for 1 year.
  Experiment Group 2: Patients underwent once RIPC 4 hours before surgery, and then normal medical procedures were performed with no additional intervention.
  Control group: Patients did not receive any additional intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): Routine treatment + interventions:The patient underwent one RIPC (Four five-minute cycles of upper limb ischaemia and Four five-minute pauses using a blood pressure cuff air vehicle to 200 mmHg) before surgery, then normal surgery, and RIPC was performed on the second day and Once RIPC/day after CABG for one year.
  Interventions: Other: remote ischemic preconditioning （RIPC）
- Experimental Group 2 (Experimental): Routine treatment + interventions:Patients underwent a RIPC before surgery, and then normal medical procedures were performed with no additional intervention.
  Interventions: Other: remote ischemic preconditioning （RIPC）
- Control group (No Intervention): routine treatment, no RIPC

INTERVENTIONS:
Other: remote ischemic preconditioning （RIPC） — Four five-minute cycles of upper limb ischaemia and Four five-minute pauses using a blood pressure cuff inflated to 200 mmHg.
  Arms: Experimental Group 1; Experimental Group 2

SUMMARY:
Remote Ischemic preconditioning (RIPC) has been reported to improve myocardial microcirculation, promote collateral circulation recruitment, and improve myocardial perfusion in patients.Two large randomized controlled trials demonstrated a perioperative cardioprotective effect of RIPC (reduced troponin levels), but did not find that a single preoperative RIPC improved long-term outcomes of coronary artery bypass grafting(CABG).The effect of a single RIPC before CABG may be too short. This study aims to investigate whether long-term RIPC improved myocardial perfusion in patients 3 months and 6 months after CABG surgery , and to detect changes in blood vascular endothelial growth factor, Nitrc Oxide, adenosine，and Endothelin-1, and to observe MACCE event rates at 12 months.

DETAILED DESCRIPTION:
A total of 210 patients were randomly divided into three groups according to the inclusion and exclusion criteria, with 70 patients in each group.

Experimental Group 1:

The patient underwent one RIPC (Four five-minute cycles of upper limb ischaemia and Four five-minute pauses using a blood pressure cuff air vehicle to 200 mmHg) 1 hours before surgery, then normal surgery, and RIPC was performed on the second day after surgery and every day after surgery, which lasted for 1 year.

Experiment Group 2:

Patients underwent once RIPC 1 hours before surgery, and then normal medical procedures were performed with no additional intervention.

Control group:

Patients did not receive any additional intervention. All patients were evaluated in three ways. First: 7days and 3 months after surgery , the quantitative examination of myocardial blood flow was conducted to observe the improvement of myocardial blood perfusion.

Second: The changes in the concentrations of vascular colorectal growth factor, Nitrc Oxide, adenosine, and endothelin-1.

Third, patients were evaluated for 6 months and 12months MACCE incidence (cardiovascular death, Nonfatal myocardial infarction, unplanned revascularization, and stroke).

ELIGIBILITY:
Inclusion Criteria:

* Three coronary artery lesions, CABG surgery was planned

Exclusion Criteria:

* The patients could not tolerate ripc;
* peripheral vascular disease affecting upper limbs
* Acute myocardial infarction complicated with cardiogenic shock，in recent 30 days,
* Emergency cases
* Severe structural heart disease and severe arrhythmia ；
* The uncontrolled systolic blood pressure and diastolic blood pressure of severe hypertension were 180 mmHg and 120 mmHg respectively;
* Severe liver, renal and pulmonary disease
* Mental disorder can't cooperate;
* Inability to give informed consent；
* Patients on glibenclamide or nicorandil, as these medications may interfere with RIC
* pregnant;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of MBF by SPECT | 3 months
  Myocardial perfusion was evaluated by Single Photon Emission Computed Tomography(SPECT): myocardial blood flow(MBF)
Change of MPR by SPECT | 3 months
  Myocardial perfusion was evaluated by Single Photon Emission Computed Tomography(SPECT): myocardial perfusion reserve(MPR)
Change of MBF by CE | 3 months
  Myocardial perfusion was evaluated by contrast echocardiography(CE): myocardial blood flow(MBF)
Change of MPR by CE | 3 months
  Myocardial perfusion was evaluated by contrast echocardiography(CE): myocardial perfusion reserve(MPR)

SECONDARY OUTCOMES:
MBF by SPECT | 1 weeks
  Myocardial perfusion was evaluated by Single Photon Emission Computed Tomography(SPECT): myocardial blood flow(MBF)
MPR by SPECT | 1 weeks
  Myocardial perfusion was evaluated by Single Photon Emission Computed Tomography(SPECT): myocardial perfusion reserve(MPR)
MBF by CE | 1 weeks
  Myocardial perfusion was evaluated by contrast echocardiography(CE): myocardial blood flow(MBF)
MPR by CE | 1 weeks
  Myocardial perfusion was evaluated by contrast echocardiography(CE): and myocardial perfusion reserve(MPR)
Rate of major adverse cardiovascular and cerebrovascular events | 12 months
  Cardiovascular death, non-fatal acute myocardial infarction, revascularization, stroke
Rate of major adverse cardiovascular and cerebrovascular events | 6 months
  Cardiovascular death, non-fatal acute myocardial infarction, revascularization, stroke
Concentration of VEGF | -1days，1 weeks，3months post surgery
  Blood vascular colorectal growth factor
Concentration of NO | -1days，1 weeks，3months post surgery
  Blood Nitrc Oxide
Concentration of BK | -1days，1 weeks，3months post surgery
  Blood bradykinin
Concentration of ET-1 | -1days，1 weeks，3months post surgery
  Blood endothelin-1
Concentration of adenosine | -1days，1 weeks，3months post surgery
  Blood adenosine
Concentration of troponin | Before surgery and after surgery
  Blood troponin
6 minute Walk Test | 1 weeks, 3/6/9 and 12 months post surgery
  6 minute Walk Test
Seattle angina questionnaire score | 1 weeks, 3/6/9 and 12 months post surgery
  Including the limited degree of physical activity, stable state of angina pectoris, angina attack frequency, treatment satisfaction, disease recognition and recognition of 5 dimensions.
Change of LVEF by SPECT | 1 weeks, 3 months,6 months
  left ventricular ejection fraction was evaluated by Single Photon Emission Computed Tomography(SPECT):

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, Ph.D, Principal Investigator — Fuwai central China cardiovascular hospotial; Zhaoyun Cheng, Ph.D, Principal Investigator — Fuwai central China cardiovascular hospotial
Locations (1):
- Fuwai central China cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
One year after the end of the trial, other outside investigators could access the original data on reasonable requests

REFERENCES:
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Background] Lau JK, Roy P, Javadzadegan A, Moshfegh A, Fearon WF, Ng M, Lowe H, Brieger D, Kritharides L, Yong AS. Remote Ischemic Preconditioning Acutely Improves Coronary Microcirculatory Function. J Am Heart Assoc. 2018 Oct 2;7(19):e009058. doi: 10.1161/JAHA.118.009058. PMID 30371329
- [Background] Meybohm P, Bein B, Brosteanu O, Cremer J, Gruenewald M, Stoppe C, Coburn M, Schaelte G, Boning A, Niemann B, Roesner J, Kletzin F, Strouhal U, Reyher C, Laufenberg-Feldmann R, Ferner M, Brandes IF, Bauer M, Stehr SN, Kortgen A, Wittmann M, Baumgarten G, Meyer-Treschan T, Kienbaum P, Heringlake M, Schon J, Sander M, Treskatsch S, Smul T, Wolwender E, Schilling T, Fuernau G, Hasenclever D, Zacharowski K; RIPHeart Study Collaborators. A Multicenter Trial of Remote Ischemic Preconditioning for Heart Surgery. N Engl J Med. 2015 Oct 8;373(15):1397-407. doi: 10.1056/NEJMoa1413579. Epub 2015 Oct 5. PMID 26436208
- [Background] Hausenloy DJ, Candilio L, Evans R, Ariti C, Jenkins DP, Kolvekar S, Knight R, Kunst G, Laing C, Nicholas J, Pepper J, Robertson S, Xenou M, Clayton T, Yellon DM; ERICCA Trial Investigators. Remote Ischemic Preconditioning and Outcomes of Cardiac Surgery. N Engl J Med. 2015 Oct 8;373(15):1408-17. doi: 10.1056/NEJMoa1413534. Epub 2015 Oct 5. PMID 26436207